CLINICAL TRIAL: NCT01634607
Title: Bone Health and Vitamin D Status in Thai HIV-1 Infected and Uninfected Adults (A Substudy of TNT-HIV 003: Trends of Morbidity and Mortality Among Thai HIV-infected and HIV-uninfected Patients: a Five-year Prospective Cohort Study)
Brief Title: Bone Health and Vitamin D Status
Acronym: BHVD
Status: Completed | Type: Observational
Sponsor: Thai Red Cross AIDS Research Centre (Other)
Collaborators: ViiV Healthcare (Industry); HIV Netherlands Australia Thailand Research Collaboration (Network); Bamrasnaradura Infectious Diseases Institute (Other Government); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Sponsor
Other Study IDs: TNT-HIV 003.1
Record Dates: First submitted 2012-07-02; First posted 2012-07-06 (Estimated); Last update posted 2023-02-17 (Actual); Status verified 2021-10

CONDITIONS: Osteopenia; Vitamin D Deficiency; HIV Infection
Keywords: osteopenia; vitamin D deficiency; HIV-infected patients; bone health; Bone mineral density (BMD); HIV-uninfected patients; effects of TDF on the patients' bone
MeSH Terms: conditions — Bone Diseases, Metabolic; Vitamin D Deficiency; HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- HIV uninfected: HIV negative patients
- HIV-infected, HAART naïve, high CD4 count: HIV positive patients with high CD4 and not on HIV treatment
- HIV-infected with planned to start HAART group: HIV positive patients who will start HIV treatment

SUMMARY:
This study will compare and assess the prevalence of osteopenia and vitamin D deficiency as well as effects of TDF on the patients' bone among HIV positive and negative patients.

DETAILED DESCRIPTION:
To determine the prevalence of osteopenia and vitamin D deficiency in HIV-1 infected, HAART naive Thai patients compared to HIV-1 uninfected Thai participants. Furthermore, to determine the change in BMD after twelve months in HIV-1 infected Thai patients on a TDF-based HAART regimen compared to patients on a non-TDF containing regimen.

ELIGIBILITY:
Inclusion Criteria:

* HIV uninfected:

  * HIV negative confirmed by HIV testing
  * Age 30 years and older
  * Thai nationality
  * Signed informed consent form for the study
* HIV-infected, HAART naïve:

  * Recorded HIV infection
  * Age 30 years and older
  * Thai nationality
  * Signed informed consent form for the study
* HIV-infected, HAART group:

  * Recorded HIV infection
  * Age 30 years and older
  * Thai nationality
  * HAART naïve at baseline, planned to start HAART within 90 days. Past exposure to antiretroviral therapy during pregnancy for the prevention of mother to child transmission of HIV ≥ 3 months prior to screening will be allowed
  * Signed informed consent form for the study

Exclusion Criteria:

* HIV uninfected

  * Currently pregnant or lactating
  * Recent hospitalization
  * Use of anticonvulsants, steroids or vitamin D supplements
* HIV-infected, HAART naïve

  * CD4 < 350
  * Currently pregnant/lactating
  * Recent hospitalization
  * Signs of wasting
  * Use of anticonvulsants, steroids or vitamin D supplements
* HIV-infected, HAART group:

  * Prior antiretroviral therapy use
  * Currently pregnant/lactating
  * Recent hospitalization
  * Signs of wasting
  * Active opportunistic infection
  * Use of anticonvulsants, steroids or vitamin D supplements

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All participants are from the Anonymous Clinic of the Thai Red Cross AIDS Research Centre (TRC-ARC, the HIV Netherlands Australia Thailand Research Collaboration (HIVNAT) and Queen Savang Vadhana Memorial Hospital (QSV).
Sampling Method: Probability Sample
Enrollment: 235 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2023-02-16 (Actual)

PRIMARY OUTCOMES:
osteopenia | 60 months
  development of osteopenia
vitamin D deficiency | 60 months
  development of vitamin D deficiency
BMD | 1 year
  changes of BMD

CONTACTS AND LOCATIONS:
Overall Officials: Praphan Phanuphak, MD, Principal Investigator — The Thai Red Cross AIDS Research Centre
Locations (1):
- The Thai Red Cross AIDS Research Centre, Pathum Wan, Bangkok, Thailand

REFERENCES:
- [Derived] Han WM, Wattanachanya L, Apornpong T, Jantrapakde J, Avihingsanon A, Kerr SJ, Teeratakulpisarn N, Jadwattanakul T, Chaiwatanarat T, Buranasupkajorn P, Ramautarsing R, Phanuphak N, Sunthornyothin S, Ruxrungtham K, Phanuphak P; TNT 003.1 study team. Bone mineral density changes among people living with HIV who have started with TDF-containing regimen: A five-year prospective study. PLoS One. 2020 Mar 25;15(3):e0230368. doi: 10.1371/journal.pone.0230368. eCollection 2020. PMID 32210458